CLINICAL TRIAL: NCT06526728
Title: Hyperbaric Oxygen Therapy in HAMstring Injury (HOTHAM) Trial
Acronym: HOTHAM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: JL Tol (Other)
Responsible Party: Sponsor-Investigator, JL Tol, Professor of Sports Medicine, Principal investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024.0395
Record Dates: First submitted 2024-07-18; First posted 2024-07-30 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Hamstring Injury
MeSH Terms: interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: 50 study participants will be treated with seven once-daily sessions of hyperbaric oxygen therapy following hamstring injury.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): Participants will be subjected to seven once-daily sessions of hyperbaric oxygen therapy.
  Generic Name: Oxygen Dosage: 100% Frequency: Once-daily Duration per treatment session: 115-120 minutes
  Interventions: Drug: Hyperbaric oxygen

INTERVENTIONS:
Drug: Hyperbaric oxygen — Participants will be subjected to seven once-daily sessions of hyperbaric oxygen therapy. Each session will last 115-120 minutes whereby the chambre will be pressurized to 2.4 ATA during which participants will breathe 100% (pure) oxygen.

SUMMARY:
The goal of this study is to learn if Hyperbaric Oxygen Therapy is able to accelerate and improve muscle healing following an acute hamstring injury. The main questions it aims to answer are:

1. Does Hyperbaric Oxygen Therapy accelerates the time needed to return to play/-duty following hamstring injury.
2. Does Hyperbaric Oxygen Therapy decrease the amount of reinjuries within 1 year following Return to play/-duty? Besides these questions this study will clinically and radiologically evaluate the healing process over time as well as the occurrence of (serious) adverse events.

DETAILED DESCRIPTION:
Trial objectives and endpoints Primary objective(s) Endpoint for the primary objective

To Compare the time needed to return to play (RTP) or -full unrestricted duty (RTD) after seven daily sessions of HBOT to a historical control group (standard care). • Time needed to return to play (days) / time needed to return to full unrestricted duty (days) defined as:

* RTP: Number of days from initial injury until the athlete is cleared to resume full unrestricted training
* RTP: Number of days from initial injury until soldier is cleared to resume full unrestricted (physical) duty activities.

Secondary objective(s), if applicable Endpoint(s) for secondary objectives Clinically assess the hamstring injury over time (Baseline, week 2 and at RTP/RTD) • Patient reported hamstring scores: Tenger activity score, Functional Assessment scale for acute hamstring injuries and psychological readiness.

* Maximum and mean pain scores (0-10) assessed with the visual analog scale, at injury, at rest and during sprinting.
* Physical examination including:

  * Palpation: Location and dimension of painful area/lesion, presence of hematoma or -swelling
  * Pain with isometric contraction against resistance
  * Hamstring flexibility tests: Passive straight leg raise, Active knee extension test.
  * Hamstring isokinetic strength (Hand hold dynamometer) Investigate MRI changes over time (Baseline, week 2)
* MRI derived parameters: Aspect of the injury on T1 and T2-weighted images scored by a radiologist using a standardized form.

Registration of re-injury rates at 2- and 12 months following initial injury • Number of re-injury at -2 and 12 months following initial injury

Assess safety of HBOT in patients with hamstring injury

• Number of AE- and SAE from signing of informed consent to 1 week following last HBOT session.

Trial design Open-label, prospective study with matched historical control cases as comparators (case-control) where participants are treated with seven daily sessions of hyperbaric oxygen therapy followed by one year of electronic follow-up.

Trial population

The trial population will consist of 50 adult (≥18 years old) athletes and military personnel with a recent (≤7 days) clinical diagnosis of an acute hamstring injury, defined as:

* Anamnestic acute injury
* Anamnestic pain in the posterior thigh
* Localized pain during palpation of the hamstring muscle
* Localized pain during passive straight leg raise
* Increased pain during isometric contraction of the hamstring muscles. Participants will not be eligible to participate in the study if they: are not capable of doing an active exercise program, have no intention to return to full sporting or duty activities, the injury is caused by extrinsic trauma, they have a chronic or recent (<2 months) hamstring injury, the injury is a complete proximal tendon avulsion, there are other injuries inhibiting recovery or if there are contra-indications for MRI or HBOT.

Interventions:

Following inclusion patients will be treated with seven daily sessions of HBOT. During this treatment patients are placed in a hyperbaric chamber in which 100% (pure) medicinal oxygen is breathed via a built-in breathing mask at a pressure of 2.4 times atmospheric pressure (equal to diving at a depth of 14 meters) for 90 min, including three 5 min 'air breaks' during which patients breathe air instead of oxygen. This treatment regime is standard within the AUMC and thus remains within the oxygen toxicity and non-decompression limits. .

On three occasions (baseline and week 2 and at RTP/RTD) participants will undergo physical examination. On two occasions (baseline and week 2) an MRI scan of the injured leg will be made. Participants will be monitored for the occurrence of re-injury at 2 and 12 months following return to sport or -unrestricted duty

ELIGIBILITY:
Inclusion Criteria:

* The participant is male or female, of any ethnic origin
* The participant is between 18 and 65 years old
* The participant has a clinical diagnosis of an acute hamstring injury ≤7 days old, defined as:

  * Anamnestic acute injury
  * Anamnestic pain in the posterior thigh
  * Localized pain during palpation of hamstring muscle
  * Localized pain during passive straight leg raise
  * Increased pain during isometric contraction
* The participant is able to start of HBOT treatment ≤7 days)

Exclusion Criteria:

* The participant is not capable of doing an active exercise program.
* The participant does not have the intention to full sporting activity or duty activities;
* The cause of the hamstring injury is an extrinsic trauma on the posterior thigh;
* The participant has a chronic hamstring injury >2 months, defined as recurrent pain or tenderness of the hamstring;
* The current injury is a re-injury ≤2months after RTP/RTD after acute ipsilateral hamstring injury;
* Clinical suspicion of a complete proximal tendon avulsions;
* Presence of other concurrent injuries inhibiting rehabilitation;
* The participant is not able to give informed consent;
* There are contra-indications for MRI: Pacemaker, pregnancy and claustrophobia
* There are contra-indications for HBOT:

  * Smoking or quit smoking <3 months prior to injury;
  * A previous spontaneous pneumothorax.
  * Implantation of ICD or PM not compatible with hyperbaric pressure
  * Current or recent (<6 months) use of cytostatics
  * Unable to perform a Valsalva manoeuvre to pressurize the middle ear (pre-existent ear-nose-throat complaints or a current upper airway infection).
  * Pregnancy
  * Claustrophobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Time to return to full unrestricted play / time to return to full unrestricted duty. | From date of inclusion until the date of progresion to return to full unrestricted play or -duty. Assessed to up to 1 year
  Number of days from initial injury until the athlete is cleard to resume full unrestricted training / Number of days from initial injury until soldier is cleared to resume full unrestricted (physical) duty activities.

SECONDARY OUTCOMES:
Re-injury registration | 2- and 12 months following injury
  Number of re-injuries
Clinical assessment | Baseline, week 2 and at return to full restricted play/-duty (assessed up to 1 year following injury)
  Clinically assess the hamstring injury over time (Patient reported hamstring scores, Pain scores), physical assessment (palpation, flexibility and isometric strength testing).
Radiologic assessment | Baseline and week 2
  Radiologic assessment of the hamstring injury over time using MRI derived parameters: Aspect of the injury on MRI images by a radiologist.
Adverse events | Baseline up until 1 week following last treatment session.
  Number of AE-and SAE's

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
IPD will not be made pubicly available but can be obtained upon request at the study's sponsor. For data reuse, a Data Sharing Agreement will be set up .